CLINICAL TRIAL: NCT06166576
Title: An Open-label, Prospective, Multi-center Clinical Trial to Evaluate the Efficacy and Safety of Ablative Radioembolization Using Yttrium-90 Glass Microspheres in Patients With Locally-advanced Hepatocellular Carcinoma
Brief Title: Radioembolization as a Spearhead Treatment of Hepatocellular Carcinoma With Localized Portal Vein Tumor Thrombosis
Acronym: RESOLVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Woo Choi, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-2306-207-1446
Record Dates: First submitted 2023-11-30; First posted 2023-12-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Radioembolization; Portal vein tumor thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radioembolization (Experimental): Hepatocellular carcinoma with localized portal vein tumor thrombosis (Vp1-Vp3) will be treated by ablative radioembolization using TheraSphere (Boston Scientific) glass microspheres
  Interventions: Procedure: Ablative radioembolization

INTERVENTIONS:
Procedure: Ablative radioembolization — The interventional radiologist utilizes a pre-test with 99mTc-MAA SPECT-CT and cone-beam CT for procedural planning. For tumors confined to a single segment, the treatment area is planned to receive a radiation dose of over 400 Gy using the single-compartment MIRD technique. For tumors extending beyond a single segment, the multi-compartment MIRD technique is used to plan a radiation dose of 700 Gy (± 20%) to the tumor. The upper limit for the estimated lung dose is set at 25 Gy, and the upper limit for the perfused non-tumoral liver dose is 250 Gy. In cases where tumors extending beyond a single segment cannot receive the planned dose of 700 Gy (± 20%) due to limits on lung or normal liver dose, the plan is adjusted to deliver the maximum dose to the tumor within the permissible range for lung and normal liver doses. Radioembolization is typically performed in a single session, and any methods not mentioned here should follow the instructions for use of TheraSphere.

SUMMARY:
The RESOLVE trial, an open-label, single-arm, multi-center study, aims to assess the efficacy and safety of ablative radioembolization using TheraSphere Yttrium-90 microspheres. This trial specifically targets patients diagnosed with hepatocellular carcinoma accompanied by localized portal vein tumor thrombosis (Vp1-Vp3) and who maintain good liver function.

DETAILED DESCRIPTION:
Patients diagnosed with unilobar hepatocellular carcinoma and localized portal vein tumor thrombosis (Vp1-Vp3), who also exhibit good liver function, will undergo ablative radioembolization with a dose exceeding 205 Gy to the tumor using TheraSphere glass microspheres. These patients will be monitored over a two-year period to evaluate their clinical course, treatment outcomes, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and over
2. Patients diagnosed with unilobar hepatocellular carcinoma, either histologically and/or radiologically (LI-RADS 4 or 5)
3. Patients with at least one measurable lesion greater than 10 mm on dynamic contrast-enhanced CT or MRI
4. Patients with localized portal vein invasion limited in one lobe (Vp1-3) on dynamic contrast-enhanced CT or MRI
5. Patients with no extrahepatic metastasis on lung CT and contrast-enhanced abdominal CT or MRI
6. Patients with no prior treatment for liver cancer
7. Child-Pugh class A
8. Eastern Cooperative Oncology Group (ECOG) performance status of 1 or less
9. Patients without serious dysfunction of major organs, as indicated by blood tests conducted within one month of study enrollment

   1. Leukocytes ≥ 2,500/µL and ≤ 12,000/µL
   2. Absolute neutrophil count ≥ 1,500/mm^3
   3. Hemoglobin ≥ 8.0 g/dL (transfusions allowed to meet this criterion)
   4. Total bilirubin ≤ 3.0 mg/dL
   5. Platelets ≥ 50,000/µL
   6. For patients not on anticoagulants, INR ≤ 2.0
   7. AST ≤ 200 IU/L (i.e., ≤ 5X upper normal limit)
   8. ALT ≤ 200 IU/L (i.e., ≤ 5X upper normal limit)
   9. ALP ≤ 575 IU/L (i.e., ≤ 5X upper normal limit)
   10. Creatinine ≤ 2.0 mg/dL
10. Patients with a life expectancy of more than 3 months
11. Patients who have fully understood the clinical trial and given written consent
12. Female patients of childbearing age confirmed not to be pregnant

Exclusion Criteria:

1. Patients unsuitable for ablative radioembolization as per the pre-test with macro-aggregated albumin labeled with technetium-99 (99mTc-MAA) for radioembolization.

   1. Cases where, according to multi-compartment Medical Internal Radiation Dose method, delivering 205 Gy of radiation to the tumor exceeds an estimated lung dose of 25 Gy.
   2. Cases with severe hepatic artery-portal vein shunting leading to expected irradiation of the non-tumorous opposite lobe.
2. Patients whose volume of non-tumorous liver not included in the treatment area is less than 30% of the total non-tumorous liver volume.
3. Patients with hepatic vein or bile duct invasion as seen on dynamic contrast-enhanced CT or MRI.
4. Patients scheduled to use immunotherapy regardless of the response to radioembolization.
5. Patients who had active cancer within two years prior to joining the clinical trial.
6. Patients who have undergone surgery or procedures related to the bile duct.
7. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time of treatment up to participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)

SECONDARY OUTCOMES:
Objective response rate according to mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Duration of response according to mRECIST | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
2-year restricted mean duration of response according to localized mRECIST and mRECIST | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or 24 months after the initial treatment
Complete response rate according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Duration of complete response according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
2-year restricted mean DoCR (RMDoCR) according to localized mRECIST and mRECIST | Time of complete response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or 24 months after the initial treatment
Best response within 2-years according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time to best response according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time to progression according to localized mRECIST and mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
2-year restricted mean survival time of overall survival | Time of treatment up to participant's death, opposition to data collection, lost to follow-up, or 24 months the initial treatment
Progression-free survival | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Hepatic progression-free survival | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Pathological necrosis rate (%) after curative resection or liver transplantation | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Time to subsequent HCC treatment | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Reason for subsequent HCC treatment | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Rate for conversion to curative resection and liver transplantation | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
Adverse event and serious adverse event | Time of treatment up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
  Common Terminology Criteria for Adverse Events v5.0
Changes in Child-Pugh class | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
Changes in ALBI (albumin-bilirubin) grade | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
Changes in MELD (Model for end-stage liver disease) score | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
Changes in ECOG (Eastern Cooperative Oncology Group) performance status scale | Baseline up to 90 days after the initial treatment or subsequent anticancer treatment, whichever comes first
  0 (fully active) to 5 (dead)
Objective response rate according to localized mRECIST | Time of treatment up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The number of patients with partial or complete response as the best local response divided by the total number of participants
Duration of response according to localized mRECIST | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (24 months after the last patient is enrolled)
  The time from first documentation of partial or complete response to the first documentation of progressive disease, death due to any cause, or receipt of subsequent anticancer treatment, whichever comes first

OTHER OUTCOMES:
Pre-treatment dosimetry based on 99mTc-MAA SPECT-CT | Baseline
Post-treatment dosimetry based on Y90 PET-CT | Within two days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Choi, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - National Cancer Center, Ilsan, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JW, Kim GM, Hyun D, Jang MJ, Kim HC. Radioembolization as a Spearhead Treatment of Hepatocellular Carcinoma with Localized Portal Vein Tumor Thrombosis (RESOLVE): Protocol for an Open-label, Multi-center, Single-arm Trial. Cardiovasc Intervent Radiol. 2025 Mar;48(3):398-404. doi: 10.1007/s00270-024-03935-2. Epub 2025 Feb 13. PMID 39948248